CLINICAL TRIAL: NCT00289107
Title: Multi-center, Prospective, Clinical Evaluation of the P.F.C.® Sigma™ Rotating Platform Cruciate Substituting vs P.F.C.® Sigma™ Cruciate Substituting Knee Primary Cases
Brief Title: Randomized Fixed Bearing vs Mobile Bearing Cruciate Substituting TKA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DePuy Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SRP-3
Record Dates: First submitted 2006-02-07; First posted 2006-02-09 (Estimated); Results first posted 2010-12-10 (Estimated); Last update posted 2023-05-03 (Actual); Status verified 2023-03

CONDITIONS: Osteoarthritis; Rheumatoid Arthritis; Other Inflammatory Arthritis; Post-Traumatic Arthritis; Juvenile Rheumatoid Arthritis; Avascular Necrosis
Keywords: Total Knee Replacement; Knee Prosthesis
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid; Arthritis, Juvenile; Osteonecrosis | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): P.F.C.® Sigma™ Rotating Platform Cruciate Substituting Knee System
  Interventions: Device: Total Knee Arthroplasty
- 2 (Active Comparator): P.F.C.® Sigma™ Fixed Cruciate Substituting Knee System
  Interventions: Device: Total knee replacement

INTERVENTIONS:
Device: Total Knee Arthroplasty — Rotating Platform (RP) Cruciate Substituting Knee System
  Other Names: P.F.C.® Sigma™ RP Cruciate Substituting Knee System
  Arms: 1
Device: Total knee replacement — Fixed Cruciate Substituting Knee System
  Other Names: P.F.C.® Sigma™ Fixed Cruciate Substituting Knee System
  Arms: 2

SUMMARY:
The study will evaluate the clinical performance of the rotating platform and fixed bearing implants through patient questionnaires, outcomes scoring and radiographic assessment.

DETAILED DESCRIPTION:
The study will evaluate the clinical performance of rotating platform and fixed bearing cruciate ligament substituting implants by obtaining a series of primary TKAS. Patients will receive either the P.F.C.® Sigma™ Rotating Platform Cruciate Substituting Knee System or P.F.C.® Sigma™ Fixed Cruciate Substituting Knee System and assignment is randomized.

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis
* Rheumatoid arthritis
* Other inflammatory arthritis
* Avascular necrosis (AVN) of bone
* Post-Traumatic Arthritis
* Juvenile Rheumatoid Arthritis

Exclusion Criteria:

* History of recent/active joint sepsis.
* Charcot neuropathy.
* Psycho-social disorders that would limit rehabilitation.
* Greater than 75 years of age at the time of surgery.
* Prior ipsilateral knee arthroplasty.
* Metabolic disorders of calcified tissues, such as Paget's disease.
* Severe diabetes mellitus.
* Joint replacement due to autoimmune disorders.
* Skeletal immaturity

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2001-04-01 (Actual); Primary Completion 2007-11-01 (Actual); Study Completion 2007-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tammy L O'Dell, EMT, CCRA, Study Director — DePuy Orthopaedics
Locations (3):
- United States (3):
  - Greensboro, North Carolina
  - Austin, Texas
  - Lakewood, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between April 2001 and October 2002, 106 subjects were recruited and enrolled at 3 US clinics by orthopaedic surgeons. Each study site could enroll up to 50 subjects (cohorts were re-assigned as necessary to complete enrollment in a timely manner). Recruitment was based on the inclusion and exclusion criteria in the clinical investigation plan.
Pre-assignment Details: Immediately before surgery, the implant type was determined according to the randomization schedule. Before treatment assignment, consented subjects could be excluded from the trial based on results of pre-operative clinical evaluations and/or radiographs, as per the exclusion criteria in the clinical investigation plan.
Groups:
- Rotating Platform: P.F.C.® Sigma™ Rotating Platform (RP) Cruciate Retaining Knee System has a modular polyethylene insert that is free to rotate around a central pivot point during knee motion.
- Fixed Bearing: P.F.C.® Sigma™ Fixed Cruciate Retaining Knee System implant has a modular polyethylene insert that is intraoperatively locked into position on the metal tibial base.
Period: Overall Study
Arm/Group | Rotating Platform | Fixed Bearing
Started | 77 | 72
Completed | 24 | 28
Not Completed | 53 | 44

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rotating Platform | Fixed Bearing | Total
Number analyzed (Participants) | 77 | 72 | 149
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.5 (6.3) | 65.5 (7.2) | 65.0 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 55 | 103
  Male | 29 | 17 | 46
Region of Enrollment [Count of Participants; unit: Participants]
  United States: United States | 77 | 72 | 149

OUTCOME MEASURES:

1. Primary Outcome: Knee Society Score
Description: The Knee Society Score (KSS) is comprised to two sections (each worth 100 points) for a maximum 200 points. One section is the Knee Society Clinical Score (KSCS) - points are given for pain, motion, and stability and points are deducted for flexion contracture, extension lag, and misalignment. The other section is the Knee Society Functional Score (KSFS) - points are assigned for walking distances and climbing stairs and points are deducted for use of walking aids. For each section, a score of 80-100 = excellent, 70-79 = good; 60-69 = fair; and < 60 = poor.
Time Frame: Pre-operative, 6 and 12 months and annually thereafter for at least 5 years.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Rotating Platform | Fixed Bearing
Number analyzed (Participants) | 77 | 72
Scores on a scale
  Pre-operative | 39.3 (15.8) | 37.2 (16.5)
  6 Months | 90.8 (13.8) | 89.2 (13.9)
  12 Months | 96.1 (6.6) | 93.0 (9.9)
  24 Months | 96.8 (7.6) | 96.0 (7.9)
  36 Months | 97.2 (5.2) | 94.3 (9.9)
  48 Months | 95.8 (5.9) | 93.7 (9.2)
  60 Months | 93.6 (9.0) | 93.5 (8.9)

2. Secondary Outcome: Complications
Time Frame: On-going to end of study
Reporting Status: Not Posted

3. Secondary Outcome: Revisions
Time Frame: On-going to end of study
Reporting Status: Not Posted

4. Secondary Outcome: Medical Imaging
Time Frame: Pre-operative, 6 and 12 months and annually thereafter for at least 5 years.
Reporting Status: Not Posted

5. Secondary Outcome: SF-12 Patient Outcomes
Time Frame: Pre-operative, 6 and 12 months and annually thereafter for at least 5 years.
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Rotating Platform | Fixed Bearing
Serious Adverse Events (participants affected / at risk) | 15/77 | 6/72
Other Adverse Events (participants affected / at risk) | 6/77 | 8/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rotating Platform (N=77) | Fixed Bearing (N=72)
Pulmonary Embolism (Vascular disorders) | 1 (1) | 1 (1)
GI Bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death (General disorders) | 3 (3) | 0 (0)
Manipulation under anesthesia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intraoperative medial collateral ligament injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Infection - superficial (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Adhesions (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Deep Vein Thrombosis, Pulmonary Embolism (Cardiac disorders) | 1 (1) | 0 (0)
Delayed wound healing (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Constipation/fecal impaction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Peripheral neuropathy or vascular disorder (Cardiac disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
General (General disorders) | 1 (1) | 0 (0)
Deep infection (Infections and infestations) | 1 (1) | 0 (0)
Cardiac Arrhythmia (Cardiac disorders) | 3 (3) | 0 (0)
Necrosis/wound slough (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rotating Platform (N=77) | Fixed Bearing (N=72)
Adhesions (Musculoskeletal and connective tissue disorders) | 6 (6) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less